CLINICAL TRIAL: NCT02378688
Title: A Phase II, Multicentre, Randomised, Double-Blind, Parallel Group, Placebo Controlled Study to Evaluate Safety, Tolerability and Clinical Efficacy of MT-1303 in Subjects With Moderate to Severe Active Crohn's Disease
Brief Title: Safety and Efficacy of MT-1303 in Subjects With Moderate to Severe Active Crohn's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MT-1303-E13
Record Dates: First submitted 2015-02-27; First posted 2015-03-04 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — amiselimod

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MT-1303 (Experimental)
  Interventions: Drug: MT-1303
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MT-1303
  Arms: MT-1303
Drug: Placebo
  Arms: Placebo

SUMMARY:
The primary objectives of the study are:

* To evaluate the safety and tolerability of MT-1303 in subjects with moderate to severe active Crohn's Disease（CD）
* To evaluate the clinical efficacy of MT-1303 in subjects with moderate to severe active CD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CD (involving small intestine and/or colon), confirmed by both endoscopy and histopathology at least 3 months prior to Visit 1
* Previous use of any type of corticosteroids or immunosuppressants for the treatment of CD
* Moderate to severe active CD defined by a CDAI score of ≥220 to ≤450 points at Visit 1

Exclusion Criteria:

* Diagnosis of ulcerative colitis, indeterminate colitis, pseudomembranous colitis or coeliac disease
* Enterocutaneous, abdominal or pelvic active fistulae, abscesses or fistulae likely to require surgery during the study
* GI surgery (including appendectomy) within 12 weeks prior to Visit 2 (Baseline) or has surgery planned or deemed likely to require surgery for CD during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2015-03; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who achieve a 100-point decrease from Baseline in CDAI(Crohn's Disease Activity Index) score (i.e., CDAI 100) at Visit 6 (Week 12) | 14 weeks

CONTACTS AND LOCATIONS:
Locations (11):
- Investigational site, City Name, Czechia
- Investigational site, City Name, France
- Investigational Site, City Name, Germany
- Investigational site, City Name, Hungary
- Investigational site, City Name, Israel
- Investigational site, City Name, Italy
- Investigational site, City Name, Japan
- Investigational site, City Name, Netherlands
- Investigational site, City Name, Poland
- Investigational site, City Name, Slovakia
- Investigational site, City Name, Ukraine